| sm(* YYIIII' | OBSTRUCTIVE SLEEP APNEA |
|---|---|
| A2. Principal Investigator Name: ADAM ADLER Id: 195273 Department: ANESTHESIOLOGY: BCM Center: | Phone: 832-824-5800 Fax: Email: acadler@bcm.edu Mail Stn: BCM320 |
| A3. Administrative Contact Name: KIMBERLY MAYFIELD Id: 160158 | Phone: 832-824-5800 Fax: Email: kmayfiel@bcm.edu |
| Section Ab: General Information A4. Co-Investigators | Email: kmayfiel@bcm.edu<br>Mail Stn: BCM320 |
| Name: ARVIND CHANDRAKANTAN Id: 195204 Department: ANESTHESIOLOGY: BCM Center: | Phone: 832-824-5800 Fax: Email: chandrak@bcm.edu Mail Stn: BCM320 |
| A5. Funding Source: Baylor College of Medicine (Internal Funding Only) A6a. Institution(s) where work will be performed: TCH: Texas Children's Hospital A6b. Research conducted outside of the United States: Country: Facility/Institution: Contact/Investigator: | |
| Phone Number: If documentation of assurances has not been sent to the Office of the Category: | of Research, please explain: |
| A8. Therapeutic Intent Does this trial have therapeutic intent? Not set yet | |
| A9. ClinicalTrials.gov Registration Section B: Exempt Request | |
| 3. Exempt From IRB Review Not Applicable Section C: Background Information | |
| Ventilatory suppression in children following opioid administration procedures (i.e. adenotonsillectomy). It is thought that patients we opioids, and especially in opioid naïve patients. Recent evidence may not predispose patients to increased opioid sensitivity in the do not have OSA. It is well known that OSA in children is significated vs. peripheral causation). The manifestation and etiologies are very process. The aim of this study is to identify if children with known greater incidence then in children without OSA. Section D: Purpose and Objectives | with obstructive sleep apnea (OSA) have increased sensitivity to in adults suggests that patients with moderate to severe OSA form of respiratory depression when compared with patients tha antly different from OSA in adults (e.g. gender predilection, centrally different in pediatric OSA making it a vastly different disease |
| The sole objective in this study is to evaluate if routine amounts of respiratory depression in children with documented obstructive obstructive sleep apnea Section E: Protocol Risks/Subjects | |
| <ul><li>E1. Risk Category</li><li>Category 3: Research involving greater than minimal risk and no yield generalizable knowledge about the subject's disorder or confect.</li><li>E2. Subjects</li></ul> | |
| Gender: Both Age: Child (3-12 yrs), Infant/Toddler (0-36 mos) | |
| Ethnicity: All Ethnicities Primary Language: English, Spanish | |
| Groups to be recruited will include: Asymptomatic patients with chronic conditions, healthy; Patients Which if any of the following vulnerable populations will be recruited Children /ulnerable populations require special protections. How will you ob | · |
| Indue coercion? Parents will be approached as ask to participate in the study. The can choose to avoid participation and or revoke their participation alter the care their child will receive. The risks include loss to corco-investigators collect data which will be stored only on the BCN however this risk is routinely managed by pediatric anesthesiology. | ey will be informed that this is completely voluntary and that they a transposit. Their participation or lack there of will not change of the fidentiality and we will reduce this risk by only having the PI and of the firewall. Additionally, there is a risk of apnea with all opioids |
| However this risk is routinely managed by pediatric anesthesiolog E3. Pregnant woman/fetus Will pregnant women and/or fetuses (as described in 45 CFR 46 Su No E4. Neonates | · |
| Will neonates of uncertain viability or nonviable neonates (as descri<br>No<br>E5. Children | bed in 45 CFR 46 Subpart B) be enrolled in the research? |
| Will children be enrolled in the research? Yes Section F: Design/Procedure | |
| F1. Design Select one category that most adequately describes your research: c) Pilot Discuss the research design including but not limited to such issues andomized to placebo group, use of control subjects, etc. | as: probability of group assignment, potential for subject to be |
| The Principal and/or co-investigators will identify children meetin Children's Hospital main campus. Those meeting enrollment crite. The study is a prospective randomized trial to identify the effect onclusion Criteria: | eria will be approached by the PI and or co-investigators. of opioids on children with obstructive sleep apnea |
| -Patients undergoing tonsillectomy or adenotonsillectomy at Texa Polysomnography with AHI >6 (study group) -Polysomnography Exclusion Criteria: Ages >8 years Patients requiring pre-medication Parental refusa intubation Patients with known or suspected difficult airway Obes | with AHI =0 or negative OSA 15 questionnaire (control group) I Opioid allergy/intolerance Patients requiring propofol for sity ¿ body mass index exceeding 30- (control group only) Known |
| cardiovascular disorders Known pulmonary disorders aside from Prematurity <35 weeks of gestation Personal of family history of <b>F2. Procedure</b> Patient Identification The Principal and/or co-investigators will identificated at Texas Childrens Hospital main campus. Those meeting en | asthma Patients with chronic oxygen requirement History of malignant hyperthermia Recent Illness entify children meeting enrollment criteria from the daily operative |
| list at Texas Childrens Hospital main campus. Those meeting en investigators. Control Group: -Patients requiring tonsillectomy/adenotonsillecto adenotonsillectomy for recurrent infection. Children with negative will be screened using the OSA 18 questionnaire, a validated clir Those with negative questionnaire scores will be included. | my without suspected OSA Children presenting for tonsillectomy sleep studies will be included. Those without formal sleep studie |
| Study Group: -Patients with Moderate to Severe OSA as docume be included if they have undergone formal sleep study evaluation using the apnea hypopnea index (AHI) and or the number desate OSA. Patients with AHI greater than 6 will be considered to have | ns. Stratification will be based on the polysomnography testing uration events according to the McGill Scoring system for pediatric moderate to severe OSA and thus eligible for inclusion |
| All patients will undergo general anesthesia per the usual practic anesthesiology attending physician. Induction will be with sevoflue Endotracheal intubation using a RAE endotracheal tube will be pure Cuffed Tube = (Age / 4) + 3. Following endotracheal intubation, such continuous positive pressure. Sevoflurane will be reduced to main anesthesia machine. The patient will be allowed to establish their patients of the process of the patient will be allowed to establish their patients. | rrane+/-nitrous oxide followed by intravenous access securement<br>erformed with the size selected using the formula: Predicted Size<br>spontaneous ventilation will be maintained without the use of<br>ntain between 0.5-0.7 MAC according to the Drager Apollo<br>r respiratory equilibrium for 3 minutes following intubation on |
| 0.21% oxygen. Baseline tidal volume (TV), respiratory rate (RR) 1mcg/kg will be administrated as a bolus (usual clinical practice) following opioid administration. Apnea or desaturation <92%) will After 10 minutes,(to study a repeated dose effect) a second dose recorded for 5 minutes. Surgery will commence as usual with additional medication to be | The TV, RR, ETCO2 will be recorded, at 5 and 10 minutes be treated by assisting ventilation as required (standard practice of 1/mcg/kg will be administered with the same TV, RR, ETCO2 |
| change to standard practice will occur the research portion will be administration to calculate change from baseline (pre-opioid). roosection G: Sample Size/Data Analysis | e prospectively recording the TV, RR, ETCO2 following opioid |
| How many subjects (or specimens, or charts) will be used in this stu-<br>Local: 50 Worldwide: 50 Please indicate why you chose the sample size proposed: | |
| Our sample size is based on a recent 2019 landmark paper inve-<br>we propose to enroll 20 control patients and 30 patients with doc<br>32. Data Analysis Provide a description of your plan for data analysis. State the types<br>of proportions, regressions, analysis of variance). Which is the PRIM | umented obstructive sleep apnea of comparisons you plan (e.g. comparison of means, comparisor |
| o the primary purposes of your study? The primary outcome will be measurement of continuous variable reported as means with SD. regression analysis will be performe obstructive sleep apnea by sleep study. | es of tidal volume, respiratory rate and end tidal CO2. these will be |
| Section H: Potential Risks/Discomforts Describe and assess any potential risks/discomforts; (physical, psycseriousness of such risks: The risks include loss to confidentiality and we will reduce this risks stored only on the BCM firewall. Additionally, there is a risk of | sk by only having the PI and co-investigators collect data which w |
| pediatric anesthesiologists and encountered in nearly all anesthe There is no long term follow up or patient related efforts required Section I: Potential Benefits | |
| Describe potential benefit(s) to be gained by the individual subject a There is no planned benefit for the patient enrolled Describe potential benefit(s) to society of the planned work. the societal benefit is understanding the impact of opioids based | on obstructive sleep apnea. The risk of opioid induced respirator |
| depression can be significant and even lethal as it has been dem Do anticipated benefits outweigh potential risks? Discuss the risk-to This study is a risk category 3, moderate risk which in this case i all anesthetics and routinely managed by pediatric anesthesiolog minimized by limiting data access to those on the protocol only | -benefit ratio. s apnea. The risks to the patient is apnea which occurs in nearly |
| Section J: Consent Procedures J1. Waiver of Consent Will any portion of this research require a waiver of consent and aut NA | horization? |
| | `oneont |
| J1a. Waiver of requirement for written documentation of C Will this research require a waiver of the requirement for written doc NA | |
| Will this research require a waiver of the requirement for written doc | |
| Will this research require a waiver of the requirement for written doo NA 12. Consent Procedures Who will recruit subjects for this study? PI PI's staff Describe how research population will be identified, recruitment proparticipant and obtaining consent, steps taken to minimize the possibetail. The PI and Co-investigator will identify patients prior to the day of Participants/parents will be approached in the preoperative area | cedures, any waiting period between informing the prospective ibility of coercion or undue influence and consent procedures in for surgery that meet inclusion/exclusion criteria. for potential enrollment. The study will be explained to the |
| Will this research require a waiver of the requirement for written doo NA 12. Consent Procedures Who will recruit subjects for this study? PI PI's staff Describe how research population will be identified, recruitment proporticipant and obtaining consent, steps taken to minimize the possibetail. The PI and Co-investigator will identify patients prior to the day of the possible of the possi | cedures, any waiting period between informing the prospective ibility of coercion or undue influence and consent procedures in for potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informe |
| Will this research require a waiver of the requirement for written doc NA 12. Consent Procedures Who will recruit subjects for this study? PI PI's staff Describe how research population will be identified, recruitment proporticipant and obtaining consent, steps taken to minimize the possibetail. The PI and Co-investigator will identify patients prior to the day of Participants/parents will be approached in the preoperative area participants parent/guardian and we will explain that all care will that their participation is optional, and can be revoked at any time associated with participation. Are foreign language consent forms required for this protocol? Yes Which of the following ways will you document informed consent in Short-Form consent documents 13. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where | cedures, any waiting period between informing the prospective ibility of coercion or undue influence and consent procedures in if surgery that meet inclusion/exclusion criteria. for potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informed without penalty. They will also be informed that no cost is |
| Will this research require a waiver of the requirement for written doo NA 12. Consent Procedures Who will recruit subjects for this study? PI Pl's staff Describe how research population will be identified, recruitment proporticipant and obtaining consent, steps taken to minimize the possibetail. The PI and Co-investigator will identify patients prior to the day of Participants/parents will be approached in the preoperative area participants parent/guardian and we will explain that all care will that their participation is optional, and can be revoked at any time associated with participation. Are foreign language consent forms required for this protocol? Yes Which of the following ways will you document informed consent in Short-Form consent documents 13. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where No 14. Children Will children be enrolled in the research? Yes | cedures, any waiting period between informing the prospective ibility of coercion or undue influence and consent procedures in if surgery that meet inclusion/exclusion criteria. for potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informed without penalty. They will also be informed that no cost is |
| Mill this research require a waiver of the requirement for written doc NA 12. Consent Procedures Who will recruit subjects for this study? Pl Pl's staff Describe how research population will be identified, recruitment proparticipant and obtaining consent, steps taken to minimize the possibetail. The Pl and Co-investigator will identify patients prior to the day of Participants/parents will be approached in the preoperative area participants parent/guardian and we will explain that all care will that their participation is optional, and can be revoked at any time associated with participation. Are foreign language consent forms required for this protocol? Yes Which of the following ways will you document informed consent in Short-Form consent documents 13. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where No 14. Children Will children be enrolled in the research? Yes 15. Neonates Will non-viable neonates or neonates of uncertain viability be involve No 16. Consent Capacity - Adults who lack capacity | cedures, any waiting period between informing the prospective billity of coercion or undue influence and consent procedures in if surgery that meet inclusion/exclusion criteria. for potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informed be without penalty. They will also be informed that no cost is languages other than English? The subjects would normally have an expectation of privacy? |
| Mill this research require a waiver of the requirement for written door NA 12. Consent Procedures Who will recruit subjects for this study? PI PI's staff Describe how research population will be identified, recruitment proporticipant and obtaining consent, steps taken to minimize the possibetail. The PI and Co-investigator will identify patients prior to the day of Participants/parents will be approached in the preoperative area participants parent/guardian and we will explain that all care will that their participation is optional, and can be revoked at any time associated with participation. Are foreign language consent forms required for this protocol? Yes Which of the following ways will you document informed consent in Short-Form consent documents 13. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where No 14. Children Will children be enrolled in the research? Yes 15. Neonates Will non-viable neonates or neonates of uncertain viability be involved. No 16. Consent Capacity - Adults who lack capacity Will Adult subjects who lack the capacity to give informed consent be No 17. Prisoners Will Prisoners be enrolled in the research? | cedures, any waiting period between informing the prospective billity of coercion or undue influence and consent procedures in if surgery that meet inclusion/exclusion criteria. for potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informed be without penalty. They will also be informed that no cost is languages other than English? The subjects would normally have an expectation of privacy? |
| Will this research require a waiver of the requirement for written doo NA 12. Consent Procedures Who will recruit subjects for this study? PI Pl's staff Describe how research population will be identified, recruitment proparticipant and obtaining consent, steps taken to minimize the possibitatil. The PI and Co-investigator will identify patients prior to the day of Participants/parents will be approached in the preoperative area participants parent/guardian and we will explain that all care will that their participation is optional, and can be revoked at any time associated with participation. Are foreign language consent forms required for this protocol? Yes Which of the following ways will you document informed consent in Short-Form consent documents 13. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where No 14. Children Will children be enrolled in the research? Yes 15. Neonates Will non-viable neonates or neonates of uncertain viability be involved. No 16. Consent Capacity - Adults who lack capacity Will Adult subjects who lack the capacity to give informed consent be No 17. Prisoners Will Prisoners be enrolled in the research? No Section K: Research Related Health Information a Will research data include identifiable subject information? | cedures, any waiting period between informing the prospective bility of coercion or undue influence and consent procedures in a surgery that meet inclusion/exclusion criteria. For potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informed without penalty. They will also be informed that no cost is a languages other than English? The subjects would normally have an expectation of privacy? The ethe subjects would normally have an expectation of privacy? |
| Will this research require a waiver of the requirement for written doo NA 12. Consent Procedures Who will recruit subjects for this study? PI PI's staff Describe how research population will be identified, recruitment proporticipant and obtaining consent, steps taken to minimize the possitetail. The PI and Co-investigator will identify patients prior to the day of Participants/parents will be approached in the preoperative area participants parent/guardian and we will explain that all care will that their participation is optional, and can be revoked at any time associated with participation. Are foreign language consent forms required for this protocol? Yes Which of the following ways will you document informed consent in Short-Form consent documents 13. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where No 14. Children Will children be enrolled in the research? Yes 15. Neonates Will non-viable neonates or neonates of uncertain viability be involved. No 16. Consent Capacity - Adults who lack capacity Will Adult subjects who lack the capacity to give informed consent be No 17. Prisoners Will Prisoners be enrolled in the research? No Section K: Research Related Health Information a Will research data include identifiable subject information? NA Information from health records such as diagnoses, progress notes, NA | cedures, any waiting period between informing the prospective bility of coercion or undue influence and consent procedures in a surgery that meet inclusion/exclusion criteria. For potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informed as without penalty. They will also be informed that no cost is alanguages other than English? The subjects would normally have an expectation of privacy? The enrolled in the research? |
| Will this research require a waiver of the requirement for written doc NA 12. Consent Procedures Who will recruit subjects for this study? Pl Pl's staff Describe how research population will be identified, recruitment proparticipant and obtaining consent, steps taken to minimize the poss detail. The Pl and Co-investigator will identify patients prior to the day of Participants/parents will be approached in the preoperative area participants parent/guardian and we will explain that all care will that their participation is optional, and can be revoked at any time associated with participation. Are foreign language consent forms required for this protocol? Yes Which of the following ways will you document informed consent in Short-Form consent documents 13. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where No 14. Children Will children be enrolled in the research? Yes 15. Neonates Will non-viable neonates or neonates of uncertain viability be involved. No 16. Consent Capacity - Adults who lack capacity Will Adult subjects who lack the capacity to give informed consent be No 17. Prisoners Will Prisoners be enrolled in the research? No Section K: Research Related Health Information a Will research data include identifiable subject information? NA Anformation from health records such as diagnoses, progress notes, NA Specific information concerning alcohol abuse: NA Specific information concerning drug abuse: NA | cedures, any waiting period between informing the prospective bility of coercion or undue influence and consent procedures in a surgery that meet inclusion/exclusion criteria. For potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informed without penalty. They will also be informed that no cost is alanguages other than English? The subjects would normally have an expectation of privacy? The enrolled in the research? |
| Will this research require a waiver of the requirement for written doc NA 12. Consent Procedures Who will recruit subjects for this study? PI PI's staff Describe how research population will be identified, recruitment proparticipant and obtaining consent, steps taken to minimize the possitetail. The PI and Co-investigator will identify patients prior to the day of Participants/parents will be approached in the preoperative area participants parent/guardian and we will explain that all care will that their participation is optional, and can be revoked at any time associated with participation. Are foreign language consent forms required for this protocol? Yes Which of the following ways will you document informed consent in Short-Form consent documents 13. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where No 14. Children Will children be enrolled in the research? Yes 15. Neonates Will non-viable neonates or neonates of uncertain viability be involve No 16. Consent Capacity - Adults who lack capacity Will Adult subjects who lack the capacity to give informed consent be No 17. Prisoners Will Prisoners be enrolled in the research? No Section K: Research Related Health Information a Will research data include identifiable subject information? NA Specific information concerning alcohol abuse: NA Specific information concerning drug abuse: NA Specific information concerning drug abuse: NA Specific information concerning sickle cell anemia: NA Specific information concerning HIV: NA | cedures, any waiting period between informing the prospective bility of coercion or undue influence and consent procedures in a surgery that meet inclusion/exclusion criteria. For potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informed as without penalty. They will also be informed that no cost is alanguages other than English? The subjects would normally have an expectation of privacy? The enrolled in the research? |
| Will this research require a waiver of the requirement for written doc NA 12. Consent Procedures Who will recruit subjects for this study? PI PI's staff Describe how research population will be identified, recruitment proporticipant and obtaining consent, steps taken to minimize the possibilitial. The PI and Co-investigator will identify patients prior to the day of Participants parent/guardian and we will explain that all care will that their participation is optional, and can be revoked at any time associated with participation. Are foreign language consent forms required for this protocol? Yes Which of the following ways will you document informed consent in Short-Form consent documents 13. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where No 14. Children Will children be enrolled in the research? Yes 15. Neonates Will non-viable neonates or neonates of uncertain viability be involved No 16. Consent Capacity - Adults who lack capacity Will Adult subjects who lack the capacity to give informed consent be No 17. Prisoners Will Prisoners be enrolled in the research? No Section K: Research Related Health Information and Will research data include identifiable subject information? NA Anformation from health records such as diagnoses, progress notes, NA Specific information concerning alcohol abuse: NA Specific information concerning sickle cell anemia: NA Specific information concerning sickle cell anemia: NA Demographic information concerning sychiatry notes: NA Demographic information (name, D.O.B., age, gender, race, etc.): NA Demographic information (name, D.O.B., age, gender, race, etc.): NA Full Social Security #: NA | cedures, any waiting period between informing the prospective bility of coercion or undue influence and consent procedures in a surgery that meet inclusion/exclusion criteria. For potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informed as without penalty. They will also be informed that no cost is alanguages other than English? The subjects would normally have an expectation of privacy? The enrolled in the research? |
| Will this research require a waiver of the requirement for written doc NA 12. Consent Procedures Who will recruit subjects for this study? PI PI's staff Describe how research population will be identified, recruitment proparticipant and obtaining consent, steps taken to minimize the possibitali. The PI and Co-investigator will identify patients prior to the day of Participants parent/guardian and we will explain that all care will that their participation is optional, and can be revoked at any time associated with participation. Are foreign language consent forms required for this protocol? Yes Which of the following ways will you document informed consent in Short-Form consent documents 13. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where No 14. Children Will Children Will Children be enrolled in the research? Yes 15. Neonates Will non-viable neonates or neonates of uncertain viability be involved. No 16. Consent Capacity - Adults who lack capacity Will Adult subjects who lack the capacity to give informed consent be No 17. Prisoners Will Prisoners be enrolled in the research? No Section K: Research Related Health Information and Will research data include identifiable subject information? NA Specific information concerning alcohol abuse: NA Specific information concerning drug abuse: NA Specific information concerning drug abuse: NA Demographic information concerning psychiatry notes: NA Demographic information concerning psychiatry notes: NA Demographic information concerning psychiatry notes: NA Partial Social Security #: NA Partial Social Security #: NA Partial Social Security #: NA Partial Social Security #: NA Partial Social Security # (Last four digits): NA Partial Social Security #: NA | cedures, any waiting period between informing the prospective bility of coercion or undue influence and consent procedures in a surgery that meet inclusion/exclusion criteria. For potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informed without penalty. They will also be informed that no cost is alanguages other than English? The subjects would normally have an expectation of privacy? The enrolled in the research? |
| Will this research require a waiver of the requirement for written doc NA 12. Consent Procedures Who will recruit subjects for this study? PI PI's starff Describe how research population will be identified, recruitment proparticipant and obtaining consent, steps taken to minimize the possibetail. The PI and Co-investigator will identify patients prior to the day of Participants/parents will be approached in the preoperative area participants/parents will be approached in the preoperative area participants on is optional, and can be revoked at any time associated with participation. Are foreign language consent forms required for this protocol? Yes Which of the following ways will you document informed consent in Short-Form consent documents 13. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where No 14. Children Will children be enrolled in the research? Yes 15. Neonates Will children be enrolled in the research? Will Adult subjects who lack the capacity to give informed consent be No 17. Prisoners Will Prisoners be enrolled in the research? No Section K: Research Related Health Information a Will research data include identifiable subject information? NA Specific information concerning alcohol abuse: NA Specific information concerning global abuse: NA Specific information concerning psychiatry notes: NA Partial Social Security #: NA Partical Social Security #: NA Partical Social Security #: NA Partical Social Security #: NA Partical Social Security #: NA Partical Social Security #: NA | cedures, any waiting period between informing the prospective bility of coercion or undue influence and consent procedures in a surgery that meet inclusion/exclusion criteria. For potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informed without penalty. They will also be informed that no cost is alanguages other than English? The subjects would normally have an expectation of privacy? The enrolled in the research? |
| Will this research require a waiver of the requirement for written doc NA 12. Consent Procedures Who will recruit subjects for this study? PI PI's staff Depris staff Depris the woresearch population will be identified, recruitment properticipant and obtaining consent, steps taken to minimize the possibility. The PI and Co-investigator will identify patients prior to the day of Participants/parents will be approached in the preoperative area participants parent/guardian and we will explain that all care will that their participation is optional, and can be revoked at any time associated with participation. Whe foreign language consent forms required for this protocol? Yes Which of the following ways will you document informed consent in Short-Form consent documents 13. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where No 14. Children Will children be enrolled in the research? Yes 15. Neonates Will non-viable neonates or neonates of uncertain viability be involved. 16. Consent Capacity - Adults who lack capacity Will Adult subjects who lack the capacity to give informed consent be No 17. Prisoners Will Prisoners be enrolled in the research? No Section K: Research Related Health Information a Will research data include identifiable subject information? NA Specific information concerning alcohol abuse: NA Specific information concerning drug abuse: NA Specific information concerning by chiatry notes: NA Specific information concerning psychiatry notes: NA Demographic information (name, D.O.B., age, gender, race, etc.): NA Demographic information (name, D.O.B., age, gender, race, etc.): NA Photographs, videotapes, and/or audiotapes of you: NA Photographs, videotapes, and/or audiotapes of you: NA What is such physical research data be secured? | cedures, any waiting period between informing the prospective bility of coercion or undue influence and consent procedures in a surgery that meet inclusion/exclusion criteria. For potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informed without penalty. They will also be informed that no cost is alanguages other than English? The subjects would normally have an expectation of privacy? The enrolled in the research? |
| Will this research require a waiver of the requirement for written doc NA 12. Consent Procedures Who will recruit subjects for this study? Pl Pris staff Describe how research population will be identified, recruitment proparticipant and obtaining consent, steps taken to minimize the possetable. The Pl and Co-investigator will identify patients prior to the day or participants/parents/guardia and we will explain that all care will that their participation is optional, and can be revoked at any time associated with participation is optional, and can be revoked at any time associated with participation. We foreign language consent forms required for this protocol? Yes Which of the following ways will you document informed consent in Short-Form consent documents 33. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where No 14. Children Will children be enrolled in the research? Yes 15. Neonates Will non-viable neonates or neonates of uncertain viability be involve No 16. Consent Capacity - Adults who lack capacity Will Adult subjects who lack the capacity to give informed consent be No 17. Prisoners Will Prisoners be enrolled in the research? No Section K: Research Related Health Information a Will research data include identifiable subject information? NA Specific information concerning alcohol abuse: NA Specific information concerning drug abuse: NA Specific information concerning sickle cell anemia: NA Specific information concerning psychiatry notes: NA Demographic information concerning psychiatry notes: NA Demographic information (name, D.O.B., age, gender, race, etc.): NA Partial Social Security # (Last four digits): NA Partial Social Security # (Last four digits): NA Portographs, videotapes, and/or audiotapes of you: NA Portographs, videotapes, and/or audiotapes of you: NA What what institution will the physical research data be kept? NA NA NA How will such physical research data be secured? NA NA NA NA NA NA NA | cedures, any waiting period between informing the prospective bility of coercion or undue influence and consent procedures in a surgery that meet inclusion/exclusion criteria. For potential enrollment. The study will be explained to the se standard regardless of their participation. They will be informed that no cost is languages other than English? It the subjects would normally have an expectation of privacy? It is enrolled in the research? In a Confidentiality medications, lab or radiology findings, etc. |
| Will this research require a waiver of the requirement for written doc NA 12. Consent Procedures Who will recruit subjects for this study? PI Pris staff Describe how research population will be identified, recruitment prosenticipant and obtaining consent, steps taken to minimize the possetal. The PI and Co-investigator will identify patients prior to the day or Participants/parents will be approached in the presperalic area will that their participation is optional, and can be revoked at any time associated with participation is optional, and can be revoked at any time associated with participation is optional, and can be revoked at any time associated with participation is optional, and can be revoked at any time associated with participation. The foreign language consent forms required for this protocol? Yes Which of the following ways will you document informed consent in Short-Form consent documents 13. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where No 14. Children Will children be enrolled in the research? Yes 15. Noonates Will non-viable neonates or neonates of uncertain viability be involved No 16. Consent Capacity - Adults who lack capacity Will Adult subjects who lack the capacity to give informed consent be No 17. Prisoners Will Prisoners be enrolled in the research? No Section K: Research Related Health Information a will research data include identifiable subject information and will research data include identifiable subject information. Specific information concerning drug abuse: NA Specific information concerning alcohol abuse: NA Specific information concerning alcohol abuse: NA Specific information concerning psychiatry notes: NA Specific information concerning psychiatry notes: NA Specific information concerning psychiatry notes: NA Our moduli such physical research data be kept? NA Author of the foliopsychiatry in the secured of the physical research data be kept? NA N | cedures, any waiting period between informing the prospective bility of coercion or undue influence and consent procedures in a surgery that meet inclusion/exclusion criteria. For potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informed without penalty. They will also be informed that no cost is languages other than English? In the subjects would normally have an expectation of privacy? In the subjects would normally have an expectation of privacy? In the research? In the research? In the research? In the research? In the research provided in the research? In the research provided secured network storage of electronic research data provided secured network storage of electronic research data |
| Will characteristication of the requirement for written doe NA 12. Consent Procedures Who will recruit subjects for this study? PP Prs staff Describe how research population will be identified, recruitment proparticipant and obtaining consent, steps taken to minimize the possibetal. The PI and Co-investigator will identify patients prior to the day of participants parent/guardian and we will explain that all care will that their participations parent/guardian and we will explain that all care will that their participations, and can be revoked at any time associated with participation. Are foreign language consent forms required for this protocol? Yes Which of the following ways will you document informed consent in Short-Form consent documents 13. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where No 14. Children Will children be enrolled in the research? Yes 15. Neonates Will non-viable neonates or neonates of uncertain viability be involved to No 16. Consent Capacity - Adults who lack capacity Will Adult subjects who lack the capacity to give informed consent be No 17. Prisoners Will Prisoners be enrolled in the research? No Section K: Research Related Health Information at No Section information concerning alcohol abuse: NA Specific information concerning alcohol abuse: NA Specific information concerning sickle cell anemia: NA Specific information concerning psychiatry notes: NA Demographic information concerning psychiatry notes: NA Demographic information concerning psychiatry notes: NA Demographic information concerning psychiatry notes: NA Demographs, videotapes, and/or audiotapes of you: NA Audit institution will the physical research data be kept? NA Audit institution will the physical research data be kept? NA NA What institution will the electronic research data be kept? NA What institution will the electronic research data be kept? NA What institution will the electronic research data be kept? NA What institution will the | cedures, any waiting period between informing the prospective billity of coercion or undue influence and consent procedures in for potential enrollment. The study will be explained to the oe standard regardless of their participation. They will be informed without penalty. They will also be informed that no cost is languages other than English? In the subjects would normally have an expectation of privacy? In the subjects would normally have an expectation of privacy? In the enrolled in the research? In the medications, lab or radiology findings, etc. |
| Will this research require a waiver of the requirement for written doc NA 2. Consent Procedures Who will recruit subjects for this study? PI PI's staff Describe how research population will be identified, recruitment proparticipant and obtaining consent, steps taken to minimize the possettetil. The PI and Co-investigator will identify patients prior to the day of participants parentify under a participant parentify under the propertity are a participant parentify under the propertity of the following ways will you document informed consent in Short-Form consent documents Short-Form consent documents 3. Privacy and Intrusivenes Will the research involve observation or intrusion in situations where No 14. Children Will children be enrolled in the research? Yes 15. Neonates Will non-viable neonates or neonates of uncertain viability be involved. 16. Consent Capacity - Adults who lack capacity Will Adult subjects who lack the capacity to give informed consent by No 16. Consent Capacity - Adults who lack capacity Will research data include identifiable subject information? No 7. Prisoners Will Prisoners be enrolled in the research? No Section K: Research Related Health Information a Will research data include identifiable subject information? NA Will research data include identifiable subject information? NA Will prisoners be enrolled in the research? NA Specific information concerning drug abuse: NA NA Specific information concerning global abuse: NA Demographic information concerning global abuse: NA Demographic information concerning psychiatry notes: NA Demographs, videotapes, and/or audiotapes of you: NA Author will such physical research data be se | cedures, any walting period between informing the prospective bilty of coercion or undue influence and consent procedures in for surgery that meet inclusion/exclusion criteria. for potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informe without penalty. They will also be informed that no cost is languages other than English? In the subjects would normally have an expectation of privacy? In the subjects would normally have an expectation of privacy? In the subjects would in the research? In the research? In the research of the research of the research data or sponsor, who will have access to identifiable research data? Including PHI, sensitive, and non-sensitive data) to sponsors this study. |
| Will this research require a waiver of the requirement for written doc NA 2. Consent Procedures Who will recruit subjects for this study? PI PI's staff Describe how research population will be identified, recruitment proparticipant and obtaining consent, steps taken to minimize the possettell. The PI and Co-investigator will identify patients prior to the day or Participantsparents will be approached in the preoperative area participantsparents will be approached in the preoperative area participants parentyguardian and we will explain that all care will had their participants parentyguardian and we will explain that all care will had their participants parentyguardian and we will explain that all care will had their participants parentyguardian and we will explain that all care will massociated with participants. The PI and Co-investigation will you document informed consent in short-Form consent documents. Which of the following ways will you document informed consent in Short-Form consent documents. 13. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where No 14. Children Will children Will children be enrolled in the research? Yes 15. Neonates Will prisonete be enrolled in the research? No 16. Consent Capacity - Adults who lack capacity Will Adult subjects who lack the capacity to give informed consent by No 17. Prisoners Will Prisoners be enrolled in the research? No 18. Consent Capacity - Adults who lack capacity Will reduce the capacity of the capacity to give information? No 19. Prisoners Will Prisoners be enrolled in the research? No 19. Section K: Research Related Health Information a Will research data include identifiable subject information? No 19. Sepecific information concerning alcohol abuse: No 20. Sepecific information concerning geochic secured will be secured w | cedures, any waiting period between informing the prospective billy of coercion or undue influence and consent procedures in for groups that meet inclusion/exclusion criteria, for potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informed that no cost is languages other than English? In the subjects would normally have an expectation of privacy? In the subjects would normally have an expectation of privacy? In the subjects would in the research? In the definition of the research? In the definition of the research data or redictions. In the research data or redictions. In the research data or redictions. In the research data or sponsor, who will have access to identifiable research data? Including PHI, sensitive, and non-sensitive data) to sponsors this study, will be minimized by only using BCM/TCH behind the BCM firew investigator. |
| Will this research require a waiver of the requirement for written doc NA 2. Consent Procedures Who will recruit subjects for this study? PI PI's staff Describe how research population will be identified, recruitment proparticipant and obtaining consent, steps taken to minimize the possibility. The PI and Co-investigator will identify patients prior to the day of participants parents will be approached in the preoperative area participants. We foreign language consent forms required for this protocol? Yes Will the research involve observation or intrusion in situations where No 14. Children Will children be enrolled in the research? Yes Situation of the preoperative of the preoperative will be involved No 15. Neonates Will non-visible neonates or neonates of uncertain viability be involved No 16. Consent Capacity - Adults who lack capacity Will Adult subjects who lack the capacity to give informed consent be No 17. Prisonors Will prisoners be enrolled in the research? No Section K: Research Related Health Information? No Section K: Research Related Health Information? No Section Information concerning alcohol abuse: No Specific information concerning alcohol abuse: No Protographic information concerning psychiatry notes: No Protographic information concerning psychiatry notes: No Protographs, videotapes, and/or audiotapes of you: No Protographs, videotapes, and/or audiotapes of you: No No Protographs, videotapes, and/or audiotapes of you: No No No Protographs, v | umentation of informed consent? bedures, any waiting period between informing the prospective billy of coercion or undue influence and consent procedures in faureory that meet inclusion/sexulation criteria, for patiential envolument. The shuty will be explained to the standard reagandess of their participation. They will be informe a without penalty. They will also be informed that no cost is languages other than English? In the subjects would normally have an expectation of privacy? It is provided secured network storage of electronic research data? Including PHI, sensitive, and non-sensitive data) to sponsors This study, Will be minimized by only using BCM/TCH behind the BCM firew investigator. It is pursone (or subject) by responsible for research related to the responsible (any expert of the total dollar amount of the properties of the properties. |
| Will into research require a waiver of the requirement for written doc NA 2. Consent Procedures Who will recruit subjects for this study? PI PI's staff Describe how research population will be identified, recruitment proporticipant and obtaining consent, steps taken to minimize the possibilities. The PI and Co-investigator will identify patients prior to the day or Participants perently waive and we will explain that all care will that their participation is optional, and can be revoked at any time associated with participation. Are foreign language consent forms required for this protocol? Yes Will the research involve observation or intrusion in situations where No 13. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where No 14. Children Will children be enrolled in the research? Yes 15. Naonates Will non-viable neonates or neonates of uncertain viability be involve No 16. Consent Capacity - Adults who lack capacity Will Adult subjects who lack the capacity to give informed consent be No 17. Prisoners Will Prisoners be enrolled in the research? No Section K: Research Related Health Information a Will research data include identifiable subject information? No Section information concerning sickle cell anemia: NA Specific information concerning sickle cell anemia: NA Specific information concerning sickle cell anemia: NA Demographic information concerning psychiatry notes: NA Demographic information concerning psychiatry notes: NA Demographic information concerning psychiatry notes: NA Demographic information concerning sickle cell anemia: NA Prison Social Security # (Last four digits): NA Demographic information concerning sickle cell anemia: NA Prison Social Security # (Last four digits): NA Prison Social Security # (Last four digits): NA Prison Social Security # (Last four digits): NA Prison Social Security # (Last four digits): NA Prison Social Security # (Last four digits): NA Prison Social Security # (Last four di | umentation of informed consent? cedures, any waiting period between informing the prospective billity of coercion or undue influence and consent procedures in faureopt that meet inclusion/sexultosin criteria, for patiential envolument. The study will be explained to the standard requaless of their participation. They will be informed that no cost is languages other than English? anguages other than English? the subjects would normally have an expectation of privacy? and Confidentiality medications, lab or radiology findings, etc. sponsor, who will have access to identifiable research data? Including PHI, sensitive, and non-sensitive data) to sponsors this study, will be minimized by only using BCM/TCH behind the BCM firew meeting and the study is the study. It is be the study of |
| Will this research require a waiver of the requirement for written doc NA 2. Consent Procedures Who will recruit subjects for this study? PI PIS staff Describe how research population will be identified, recruitment por positional and obtaining consent, steps taken to minimize the possibilities. The PI and Co-investigator will tidentify patients prior to the day or Participants parentisy will be approached in the preoperative area participants parentisy will be approached in the preoperative area participants parentisy will be approached in the preoperative area participants parentisy will be approached in the preoperative area participants parentisy will pout document informed consent in the following ways will you document informed consent in Short-Form consent documents 13. Privacy and Intrusiveness Will the research involve observation or intrusion in situations where No 14. Children Will children Will children be enrolled in the research? Yes 15. Neonates Will Prisonates Will Prisonates be enrolled in the research? No 16. Consent Capacity - Adults who lack capacity Will Audit subjects who lack the capacity to give informed consent be No 17. Prisonares Will Prisoners be enrolled in the research? No Section K: Research Related Health Information a Will research data include identifiable subject information? No Prisonation from health records such as diagnoses, progress notes, Na Specific information concerning drug abuse: NA Specific information concerning psychiatry notes: NA Prisonation from health records such as diagnoses, progress notes, Na Specific information concerning psychiatry notes: NA Prisonation from the prisonation of the prison | umentation of informed consent? bedures, any waiting period between informing the prospective billy of coercion or undue influence and consent procedures in faureory that meet inclusion/sexulation criteria, for patiential envolument. The shuty will be explained to the standard reagandess of their participation. They will be informe a without penalty. They will also be informed that no cost is languages other than English? In the subjects would normally have an expectation of privacy? It is provided secured network storage of electronic research data? Including PHI, sensitive, and non-sensitive data) to sponsors This study, Will be minimized by only using BCM/TCH behind the BCM firew investigator. It is pursone (or subject) by responsible for research related to the responsible (any expert of the total dollar amount of the properties of the properties. |
| All this research require a waiver of the requirement for written doc NA 2. Consent Procedures Mino will recruit subjects for this study? Per starf Describe how research population will be identified, recruitment prosenticipant and obtaining consent, steps taken to minimize the possibility. Per land Convessigator will identify patients prior to the day. Perfoliopants/parents will be approached in the procentive area harticipants are institution and can be revoked at any time associated with participation. We foreign language consent forms required for this protocor? Yes 13. Privacy and Intrusiveness 14. Children 14. Children 15. Neonates 15. Neonates 16. | umentation of informed consent? bedures, any waiting period between intermining the prospective bility of coercion or undue influence and consent procedures in for potential enrollment. The study will be explained to the for potential enrollment. The study will be explained to the for potential enrollment. The study will be explained to the procedures in the procedure of the will be informed as without penalty. They will also be informed that no cost is languages other than English? be subjects would normally have an expectation of privacy? and in research? de enrolled in the research? and Confidentiality medications, lab or radiology findings, etc. sponsor, who will have access to identifiable research data? including PHI, sensitive, and non-sensitive data) to sponsors this study, will be minimized by only using BCM/TCH behind the BCM firew invostigator. This study, the study of the properties, during the properties, the study of the payment, paid upon completion, etc) of the payment. Subsequent to participation in this research. Please discuss, ability, employability, immigration status, patently status, subling, employability, immigration status, patently status, abolity, employability, immigration status, patently status, abolity, employability, immigration status, patently status, abolity, employability, immigration status, patently status, abolity, employability, immigration in this research. Please discuss, abolity, employability, immigration status, patently status, abolity, employability, immigration status, patently status, abolity, employability, immigration in this research. Please discuss, abolity, employability, immigration status, patently status, abolity, employability, immigration status, patently status, abolity, employability, immigration in this research. Please discuss, abolity, employability, immigration status, patently status, abolity, employability, immigration in this research. |
| Mill this research require a waiver of the requirement for written doc NA 2. Consent Procedures Who will recruit subjects for this study? PI's staff Describe how research population will be identified, recruitant processors betwin. The PI and Co-investigator will identify patients prior to the day of Participants parents will be approached in the preoperative area to the PI and Co-investigator will identify patients prior to the day of Participants parents will be approached in the preoperative area to the Participants processors and the preoperative area to the Participants of the PI and Co-investigator will identify patients prior to the day of Participants processors. The PI and Co-investigator will identify patients prior to the day of Participants processors. The PI and Co-investigator will identify patients prior to the day of Participants and the Participants. Are foreign language consent forms required for this protocor? Yes Which of the following ways will you document informed consent in Short-Form consent documents. No. Privacy and Intrusiveness Will the search involve observation or intrusion in situations where No. 14. Children Will children Will children Will children be enrolled in the research? Yes 15. Neonate Will non-value reconates or neonales of uncertain viability be involved No. 16. Consent Capacity - Adults who lack capacity Will Adult subjects who lack the capacity to give informed consent be No. No. Section K: Research Related Health Information a Will research data include identifiable subject information? No. Section From the will be recarded as a secure of the processor of the No. Privacy of the Pi and | umentation of informed consent? cedures, any waiting period between informing these prospective billty of caercion or undue influence and consent procedures in f surgery that meet inclusion/exclusion criteria. The standard regardless of their participation. They will be informed standard regardless of their participation. They will be informed that no cost is exclusive period that no cost is anguages other than English? the subjects would normally have an expectation of privacy? et a currelled in the research? a enrolled in the research? a enrolled in the research? the subjects would normally findings, etc. sponsor, who will have access to identifiable research data? including PHI. sensitive, and non-sensitive data) to sponsors this study, will be minimized by only using BCM/TCH behind the BCM firew investigator. The insurance (or subject) be responsible for research related it be responsible (surgery, device, drugs, etc). If appropriate, this study, will be minimized by only using BCM/TCH behind the BCM firew investigator. The insurance for subject) be responsible for research related it be responsible (surgery, device, drugs, etc). If appropriate, this study, will be my period to the study of the payment, paid upon completion, etc) of the payment. Subsequent to participation in this research. Please discuss, ability, employability, immigration status, paternly status, and if so, who will provide the education or counseling and under the payment. |
| All this research require a walver of the requirement for writhen doc NA. 2. Consent Procedures Who will recruit subjects for this study? PTs stall Describe how research population will be identified, recruitment procedures and obtaining consent, steps taken to minimize the possession and obtaining consent, steps taken to minimize the possession and obtaining consent break part of the the part and Co investigator will identify patients prior to the day a participants parent/guardian and we will explain that all care will that their participation is applicant, and can be revoked at any time associated with participation. We foreign language consent toms required for this protocol? Yes Who Interest to the following ways will you document informed consent in Shru-Form consent documents 33. Privacy and Intrusivoness Will the research involve observation or intrusion in situations where No 14. Children Will the research involve observation or intrusion in situations where No 15. Neonates Will include be enrolled in the research? Yes Will Adult subjects who lack the capacity to give informed consent by No 17. Prisoners Will Prisoners be enrolled in the research? No Section K: Research Related Health Information a Will research data include identifiable subject information? No Section Information concerning alcohol abuse: NA Specific information concerning globals cell anemia: NA Prisoners be enrolled in the research data be kept? NA Specific information concerning globals cell anemia: NA Prisoners information concerning psychiatry notes: NA Specific information concerning globals cell anemia: NA Prisoners information concerning psychiatry notes: NA Prisoners information concerning of the psychiatry informatio | umentation of informed consent? cedures, any waiting period between informing these prospective billy of caercion or undue influence and consent procedures in f surgery that meet inclusion-exclusion criteria. The patiental amoultment. This study will be explained to the petandard regardes of their participation. They will be informed without penalty. They will also be informed that no cost is languages other than English? the subjects would normally have an expectation of privacy? et also be unformed that no cost is entirely and the subjects would normally have an expectation of privacy? et also in research? the subjects would normally have an expectation of privacy? et allowed the research? the information of radiology findings, etc. sponsor, who will have access to identificable research data? including PHL sensitive, and non-sensitive data) to sponsors including PHL sensitive, and non-sensitive data) to sponsors this study, will be minimized by only using BCM/TCH behind the BCM firew investigator. This study. It insurance (or subject) be responsible for research related to be responsible (surgery, device, drugs, clc). If appropriate, this study, will be minimized by only using BCM/TCH behind the BCM firew investigator. It is insurance for subject) be responsible for research related to be responsible (surgery, device, drugs, clc). If appropriate, this study, will be provide the color of the payment, related to provide the color of the payment. |
| Will this research require a waiver of the requirement for written doc NA 2. Consent Procedures Who will recruit subjects for this study? PP 3 staff Describe how research population will be identified, recruitment processing and obtaining consent, sleeps taken to minimize the possibility of the processing of the proc | umentation of informed consent? coclures, any waiting period between informing the prospective billity of coercion or under influence and consent procedures in 6 surgery that meet inclusion occusion orders. for potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informe without penalty. They will also be informed that no cost is anguages other than English? the subjects would normally have an expectation of privacy? the subjects would normally have an expectation of privacy? and Confidentiality medications, lab or radiology findings, etc. the study, will be minimized by only using BCM/TCH behind the BCM firew movestigator. It is insurance (or subject) be responsible for research related be responsible (surgery, device, drugs, etc). If appropriate, the processing of the payment, paid upon completion, etc) of the payment. It is insurance (or subject) be responsible for research related be responsible (surgery, device, drugs, etc). If appropriate, this is research project, please note the total dollar amount of payment, paid upon completion, etc) of the payment. It is not in this research project, please note the total dollar amount of payment, paid upon completion, etc) of the payment. It is not if so, who will provide the education or counseling and under any special payment, paid upon completion and project please describe and if so, who will provide the education of counseling and under mily's progress purposes) |
| An internation from the research for without do NA 2. Consent Procedures The work of the receive of the requirement for without do NA 2. Consent Procedures The plant of the receive of the study? Plant at aff Beaches he were search population will be identified, recruitment properties of the study. Plant of the plant oce-investigator will identify patients prot or instance and obtaining consent, steps taken to minimize the possibility. The Plant Oce-investigator will identify patients prot or incomment and obtaining consent forms required for this protocol? Per participation is optional, and can be revoked at any time associated with participation. We foreign language consent forms required for this protocol? Yes The Plant of the tolowing ways will you document informed consent in Short-Form consent documents. An introduce the consent of the study of t | umentation of informed consent? coclures, any wairing period between informing the prospective billy of coercion or under influence and consent procedures in for potential continer. The study will be explained to the potential continer. The study will be explained to the be standard regardless of their participation. They will be informe without penalty. They will also be informed that no cost is anguages other than English? It the subjects would normally have an expectation of privacy? It the subjects would normally have an expectation of privacy? It is explained in the research? It is not research? It is not research project, please note the total dollar amount of payment, paid upon completion, etc) of the payment. It is insurance (or subject) be responsible for research related the responsible (surgery, device, drugs, etc). If appropriate, this study, will be minimized by only using BCM/TCH behind the BCM firewinessigator. It insurance (or subject) be responsible for research related the responsible (surgery, device, drugs, etc). If appropriate, this study, and it is research project, please note the total dollar amount of payment, paid upon completion, etc) of the payment. It is not research project, please note the total dollar amount of payment, paid upon completion, etc) of the payment. It is not research project, please note the total dollar amount of payment, paid upon completion, etc) of the payment. It is not research project, please note the total dollar amount of payment, paid upon completion, etc) of the payment. |
| Will be research forgete a valver of the requirement for written don'NA 2. Consent Procedures the will const subjects for this study? Pris staff Beaches now research population will be identified, recruitment prisonance, and an advantage consent, steps taxen to minimize the posterial. The Plant Ch-investigator will identify patients prior to the day or participation and obtaining consent, steps taxen to minimize the posterial. The Plant Ch-investigator will identify patients prior to the day or participation and obtaining consent, steps taxen to minimize the posterial. The Plant Ch-investigator will identify patients prior to the day or participation and the patient patient pa | umentation of informed consent? coclures, any waiting period between informing the prospective billity of coercion or under influence and consent procedures in 6 surgery that meet inclusion occusion orders. for potential enrollment. The study will be explained to the be standard regardless of their participation. They will be informe without penalty. They will also be informed that no cost is anguages other than English? the subjects would normally have an expectation of privacy? the subjects would normally have an expectation of privacy? and Confidentiality medications, lab or radiology findings, etc. the study, will be minimized by only using BCM/TCH behind the BCM firew movestigator. It is insurance (or subject) be responsible for research related be responsible (surgery, device, drugs, etc). If appropriate, the processing of the payment, paid upon completion, etc) of the payment. It is insurance (or subject) be responsible for research related be responsible (surgery, device, drugs, etc). If appropriate, this is research project, please note the total dollar amount of payment, paid upon completion, etc) of the payment. It is not in this research project, please note the total dollar amount of payment, paid upon completion, etc) of the payment. It is not if so, who will provide the education or counseling and under any special payment, paid upon completion and project please describe and if so, who will provide the education of counseling and under mily's progress purposes) |
| Note that cressorth require a walver of the requirement for written dor NA 2. Consent Procedures Thin will recent subjects for this study? Plant at at a control subjects for this study? Plant at a control subjects for this study? Plant at a control subjects for this study? Plant at a control subject for this study? Plant at a control subject for this study? Plant and Control subject for this protect prior to the day for this protect prior to the day for the protection of the day for the protection of the day for the protection of the day for the protection of the day for the protection of the control that the protection of the control that the protection of the control that the protection of the control that the protection of the control that the contro | cedures, any waiting period between informing the prospective billy of ceretron or routeness and consent procedures in fargrapy that meet industricate intension that is required to the ceretron of the study sold be explained to the between the study sold between the informed that no cost is subject to the ceretron of the study sold between the informed without penalty. They wait also be informed that no cost is languages other than English? It has subjects would normally have an expectation of privacy? It has subjects would normally have an expectation of privacy? It is enrolled in the research? It is considered that the control of the con |